CLINICAL TRIAL: NCT01494168
Title: Longitudinal Assessment of the Effect of Bariatric Surgery on Arterial Function and Blood Pressure Target Organs Damage
Brief Title: Bariatric Surgery, Arterial Stiffness and Target Organ Damage Study (BASTOD)
Acronym: BASTOD
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 8686; 2010-A01447-32 (Other: AFSSAPS)
Record Dates: First submitted 2011-11-17; First posted 2011-12-16 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension; Obesity
Keywords: Hypertension; Arterial stiffness; Obesity; Bariatric surgery
MeSH Terms: conditions — Hypertension; Obesity | interventions — Bariatric Surgery; Anastomosis, Roux-en-Y

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Bariatric surgery (Roux-en-y bypass or sleeve gastrectomy) — Bariatric surgery
  Other Names: Roux-en-y bypass; sleeve gastrectomy

SUMMARY:
Introduction:

Obesity is a major public health problem, associated with many morbidities, including metabolic and cardiovascular disease (CVD). High blood pressure (hypertension) is the most common comorbidity and one of the major risk factors for CVD and kidney failure. It has been described an almost linear relationship between body mass index (BMI) and the level of blood pressure (BP), but the mechanisms underlying this relationship are complex and incompletely understood : activation of renin-angiotensin-aldosterone and sympathetic nervous systems, alterations in systemic hemodynamics and arterial parameters; a significant correlation between overall and / or visceral obesity and arterial stiffness assessed by carotid-femoral pulse wave velocity (PWV) has been observed.

By its effectiveness in terms of magnitude and sustainability of weight loss, bariatric surgery is becoming increasingly important in the management of obesity and the prevention of its comorbidities. It reduces all-cause as well as CV mortality. Bariatric surgery allows a resolution of the metabolic syndrome (in 2 out of 3 patients) and diabetes (in 5 out of 6 patients), but its effect on blood pressure remains inconstant and transient. The reasons for this limitation and the detailed effects of bariatric surgery on hemodynamics and arterial parameters have been poorly studied. Of note, a reduction in left ventricular hypertrophy, an improvement in diastolic dysfunction and aortic distensibility assessed by ultrasound or MRI have been observed.

DETAILED DESCRIPTION:
Objective:

The study aims to (a) estimate the effects of bariatric surgery on the function of large arteries (determined non-invasively by measurement of PWV, pressure central reflection wavelength) in a population of obese grade 2 or 3, and (b) evaluate the respective role of weight loss, the change in metabolic parameters, and the decline in BP on changes in the function of large arteries and on markers of target organ alterations after surgery.

Methods:

This is a prospective longitudinal study with assessment of arterial stiffness before and after 6 and 12 months following bariatric surgery. Ninety grade 2-3 obese patients with an indication of bariatric surgery will be included. Arterial stiffness is estimated by the aortic PWV (SphygmoCor®) at baseline and after 6 and 12 months following surgery. Changes in the central pressure, wave reflection, the PA device, and markers of target organ alteration (left ventricular mass, LVM, glomerular filtration rate, GFR, urinary albumin excretion, EUA; caliber of retinal vessels as assessed by retinography) will be the secondary objectives.

To study the evolution of PWV in connection with weight loss, a linear mixed model is used based on data collected for each patient every time. Correlations between different parameters will be studied each time. Changes in secondary endpoints over time will be correlated to changes in weight, BMI, percentage loss of excess weight and blood pressure.

Expected results and their prospects:

Weight loss surgery should lead to a rapid and sustained weight loss, improved arterial function parameters (BP, arterial stiffness) and markers of target organ damage (GFR, UAE, LVM, caliber of retinal vessels).

The analysis of the relation between the metabolic / hemodynamic responses and target organ damage should enable us to identify consistent pathophysiological mechanisms, and refine our understanding of the consequences of bariatric surgery.

ELIGIBILITY:
Inclusion criteria:

* BMI > 40 kg/m2 or BMI 35-40 with major comorbidities
* Age between 18-60 years
* Obesity evolving for more than 5 years
* Failure of medical treatment
* Elimination of hormonal causes

Exclusion criteria:

* Uncontrolled hypertension (SBP > 160 mmHg and DBP> 100 mmHg).
* History of cardiovascular disease or signs of clinical atheroma: stroke, myocardial infarction and coronary heart disease (angina), peripheral arterial disease (no pulse, claudication), aortic aneurysm (anterior abdominal palpation or imaging ), carotid bruit
* Plasma creatinine > 130 micromol/L and/or proteinuria > 300 mg/24 h and/or dipstick hematuria.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: obese patient candidate for bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-12; Primary Completion 2015-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness | 6 and 12 month (plus or minus 30 days) after bariatric surgery
  Change in Arterial stiffness at 6 and 12 months(determined non-invasively by measurement of PWV, central pressure and reflection wavelength)

SECONDARY OUTCOMES:
Changes at 6 and 12 months | at 6 and 12 months
  Changes at 6 and 12 months in central pressure, wave reflection, blood pressure , and target organ damage (left ventricular mass, glomerular filtration rate, urinary albumin excretion, caliber of retinal vessels)

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Sardinoux, M.D., Principal Investigator — UH Montpellier
Locations (1):
- University Hospital, Montpellier, France